CLINICAL TRIAL: NCT04614545
Title: The Use of a Virtual Weight Management Program for Prescription of Phentermine in Patients With Overweight or Obesity Compared to Standard Face to Face Visits
Brief Title: Comparing a Virtual vs. Face to Face Weight Management Program Using Phentermine for Patients With Overweight or Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Marcio Griebeler, Staff Endocrinologist, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-948
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Results first posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Phentermine; Resistance Training

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Single-center, Parallel-group trial comparing the use of virtual visit for prescription of phentermine versus standard face-to-face visits for weight management
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Virtual Visits (Experimental): All patients will be seen face to face on visit 1. Patient will be evaluated by an obesity-medicine specialist and also by a registered dietitian and exercise physiologist via telemedicine. Subjects will be prescribed phentermine (37.5 mg po daily; dose may be reduced if not tolerated), and will choose one of two dietary programs (Mediterranean or Keto diet). Weight and vital signs will be monitored remotely and patients will receive a remote scale and a remote blood pressure cuff.
  Subjects will then initiate 3 one to one virtual visits with the obesity specialist. On each of this visit the five pillars of weight management will be discussed including nutrition, physical activity, appetite control, sleep issues, and anxiety/depression/stress. A personalized nutrition and exercise program will be developed. If felt relevant by the provider, subjects may also be referred to a mental health specialist and/or sleep clinic. All medical care will be provided virtually.
  Interventions: Drug: Phentermine 37.5 Mg; Behavioral: Dietary program; Behavioral: Exercise program
- Face to face visits (Active Comparator): All patients independently of the randomization arm will be seen face to face on visit 1. Patients will be evaluated by an obesity-medicine specialist and patient will also be seen face to face by a registered dietitian and exercise physiologist. Subjects will be prescribed phentermine (37.5 mg po daily; dose may be reduced if not tolerated). Patients will choose one of two dietary programs (Mediterranean or Keto diet). Weight and vital signs will be monitored in each of the visits.
  Subjects will then initiate 3 face to face visits with the obesity specialist provider every 4 weeks. The five pillars of weight management will be discussed including nutrition, physical activity, appetite control, sleep issues, and anxiety/depression/stress.
  The patient will be provided a personalized nutrition and exercise program and may be referred to a mental health specialist and/or sleep clinic per provider discretion. All medical care will be provided via a face-to-face manner.
  Interventions: Drug: Phentermine 37.5 Mg; Behavioral: Dietary program; Behavioral: Exercise program

INTERVENTIONS:
Drug: Phentermine 37.5 Mg — Patients will receive 37.5 mg of phentermine daily for a 12 week duration
  Other Names: Lomaira
Behavioral: Dietary program — Patients will be able to select either the Mediterranean diet or the Ketogenic diet and will work with a dietician
Behavioral: Exercise program — Patients will be provided with a personalized exercise program

SUMMARY:
This study will study the effects associated with the prescription of phentermine in a virtual setting, comparing with prescription of phentermine via a standard face-to-face visit for patients with obesity or overweight.

DETAILED DESCRIPTION:
Obesity is a major healthcare problem in the United States affecting over one-third of the population, often increasing the risk of other comorbidities like hypertension, dyslipidemia, type 2 diabetes mellitus (1) and is also associated with increased risk of all-cause mortality and cardiovascular death. Modest weight loss of 5% has been associated with improvement in obesity as well as obesity related comorbidities and quality of life. (2) The cornerstone for treatment of obesity is behavioral modification and lifestyle changes including dietary modification and physical activity. (3) Adaptive physiologic responses due to increased appetite makes it difficult to achieve weight loss with lifestyle intervention alone. Anti-obesity medications (AOM) are often required as adjuvant therapy for weight loss induction and maintenance, and have the potential to augment further weight loss. (4)

Obesity is a chronic disease that often requires chronic treatment and the use of FDA-approved medications to reduce the appetite set-point in the hypothalamus. Currently, the United States Food and Drug Administration (FDA)-approved medications include: phentermine, phentermine-topiramate (Qsymia), bupropion-naltrexone (Contrave), orlistat (Xenical, Alli) and liraglutide (Saxenda). AOMs remain underutilized and just a minority of patients receive prescription treatment due to cost of therapy, lack of insurance coverage, old requirements of frequent face-to-face visits, lack of physician training, among others. Phentermine is the most affordable and the most commonly prescribed pharmacotherapy for weight loss; however, FDA approval is only for the short-term use (90 days), and in the State of Ohio, face-to-face visits every 30 days were required until recently during the course of treatment. (5) A recent study found that in real-world practice AOMs are associated with clinically meaningful additional weight loss and phentermine therapy was associated with the most weight loss (3.7% weight loss in 12 weeks and an average of 7-12% when enhanced to our current weight management program. (6). Another study has demonstrated that phentermine is one of the most cost-effective pharmacologic weight-loss strategies. (7)

A barrier to successful weight loss is patient attrition, as often more than half of patients do not complete lifestyle-based weight loss intervention. (8) Scalable methods for the delivery of obesity treatment that encourages patient participation are needed. A potential way to improve patient participation and weight loss outcomes is through the use of virtual medical visits, remote monitoring, and e-Health. Telemedicine is a growing segment of medical field with the potential to improve access to care removing geographic barriers, extending care to home with the introduction with new technology capabilities that patients are already using on their personal lives. These new modalities have the potential to decrease costs, provide scalable and more accessibility and provide the same quality of care. Several studies have shown the utility of e-Health in the management of chronic conditions, concluding the behavioral changes can be achieved using technological innovation. (9, 10)

More recently, the emergency COVID-19 pandemic presented an unprecedented challenge to the current healthcare system, and all institutions are rapidly changing their health care delivery model and quickly adopting telemedicine and remote monitoring and very soon this type of care may become standard. Frequent visits have been shown to be effective facilitating changes in lifestyle, while also addressing psychological aspects. During the last few months, the Endocrinology and Metabolism Institute (EMI) at Cleveland Clinic has switched obesity care to essentially 90% virtual visits. In addition, the federal government and the State of Ohio recently relaxed standards for prescribing controlled substances so providers are now able to prescribe phentermine (and other anti-obesity medications) via telemedicine. If the study is able to demonstrate that a meaningful and safe weight loss can also be achieved via virtual care, this could support making current relaxed recommendations of the State of Ohio permanent, which would represent a significant shift in the current laws and would greatly benefit the care of patients suffering with obesity.

Cleveland Clinic's weight management clinic provides an ideal environment to investigate the impact of virtual weight management program for the prescribing of phentermine. The proposed trial will afford the opportunity to study the effects of a well-established weight management program associated with the prescription of phentermine in a virtual setting, comparing its effects with standard face-to-face visit. At the present time, there are no studies which have demonstrated that the use of phentermine, prescribed via telemedicine, will lead to the same outcomes in terms of weight loss. This gap in the literature needs to be rapidly answered in order to shift the current standard of weight management care from face-to-face to virtually provided care. This trial has the potential to lead to major impact on how we manage patients with obesity. If the study shows that a virtual weight management program may be as effective as face-to-face encounters for prescription of anti-obesity mediation (initially with phentermine due to feasibility) this will pave the way for future clinical trials leveraging virtual care as standard of care for management of obesity and prescription of anti-obesity medications.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* Body mass index (BMI) greater than or equal to 27 with 1 or more comorbidities (hypertension, diabetes, sleep apnea, fatty liver disease, PCOS, dyslipidemia, congestive heart failure, osteoarthritis) OR a BMI or 30 or greater
* Able to log into an online platform or have a smartphone
* Willing to join a virtual weight management program

Exclusion Criteria:

* Contraindication for use of phentermine
* Female who is pregnant, breast-feeding, or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods
* Participation in another clinical trial within 30 days of screening
* Cardiovascular disease including uncontrolled hypertension or history of arrhythmias
* Treatment with any medication with the intention of weight loss within 180 days before screening
* Use of Topiramate within 180 days of screening
* Previous history of bariatric surgery or use of minimally invasive weight loss devices

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2022-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcio Griebeler, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flegal KM, Kruszon-Moran D, Carroll MD, Fryar CD, Ogden CL. Trends in Obesity Among Adults in the United States, 2005 to 2014. JAMA. 2016 Jun 7;315(21):2284-91. doi: 10.1001/jama.2016.6458. PMID 27272580
- [Background] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ, Jordan HS, Kendall KA, Lux LJ, Mentor-Marcel R, Morgan LC, Trisolini MG, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. Circulation. 2014 Jun 24;129(25 Suppl 2):S102-38. doi: 10.1161/01.cir.0000437739.71477.ee. Epub 2013 Nov 12. No abstract available. PMID 24222017
- [Background] Bersoux S, Byun TH, Chaliki SS, Poole KG. Pharmacotherapy for obesity: What you need to know. Cleve Clin J Med. 2017 Dec;84(12):951-958. doi: 10.3949/ccjm.84a.16094. PMID 29244650
- [Background] Moroshko I, Brennan L, O'Brien P. Predictors of dropout in weight loss interventions: a systematic review of the literature. Obes Rev. 2011 Nov;12(11):912-34. doi: 10.1111/j.1467-789X.2011.00915.x. Epub 2011 Aug 5. PMID 21815990
- [Background] Wadden TA, Neiberg RH, Wing RR, Clark JM, Delahanty LM, Hill JO, Krakoff J, Otto A, Ryan DH, Vitolins MZ; Look AHEAD Research Group. Four-year weight losses in the Look AHEAD study: factors associated with long-term success. Obesity (Silver Spring). 2011 Oct;19(10):1987-98. doi: 10.1038/oby.2011.230. Epub 2011 Jul 21. PMID 21779086
- [Background] Hendricks EJ, Srisurapanont M, Schmidt SL, Haggard M, Souter S, Mitchell CL, De Marco DG, Hendricks MJ, Istratiy Y, Greenway FL. Addiction potential of phentermine prescribed during long-term treatment of obesity. Int J Obes (Lond). 2014 Feb;38(2):292-8. doi: 10.1038/ijo.2013.74. Epub 2013 May 17. PMID 23736363
- [Result] Wing RR, Lang W, Wadden TA, Safford M, Knowler WC, Bertoni AG, Hill JO, Brancati FL, Peters A, Wagenknecht L; Look AHEAD Research Group. Benefits of modest weight loss in improving cardiovascular risk factors in overweight and obese individuals with type 2 diabetes. Diabetes Care. 2011 Jul;34(7):1481-6. doi: 10.2337/dc10-2415. Epub 2011 May 18. PMID 21593294
- [Result] Apovian CM, Aronne LJ, Bessesen DH, McDonnell ME, Murad MH, Pagotto U, Ryan DH, Still CD; Endocrine Society. Pharmacological management of obesity: an endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2015 Feb;100(2):342-62. doi: 10.1210/jc.2014-3415. Epub 2015 Jan 15. PMID 25590212
- [Result] Shibuya K, Ali KF, Ji X, Milinoivh A, Bauman J, Kattan MW, Pantalone KM, Burguera B. THE BENEFIT OF SHORT-TERM WEIGHT LOSS WITH ANTI-OBESITY MEDICATIONS IN REAL-WORLD CLINICAL PRACTICE. Endocr Pract. 2019 Oct;25(10):1022-1028. doi: 10.4158/EP-2019-0081. Epub 2019 Jun 26. PMID 31241358
- [Result] Lee M, Lauren BN, Zhan T, Choi J, Klebanoff M, Abu Dayyeh B, Taveras EM, Corey K, Kaplan L, Hur C. The cost-effectiveness of pharmacotherapy and lifestyle intervention in the treatment of obesity. Obes Sci Pract. 2019 Dec 10;6(2):162-170. doi: 10.1002/osp4.390. eCollection 2020 Apr. PMID 32313674
- [Derived] Griebeler ML, Butsch WS, Rodriguez P, Lomeli L, Kampert M, Makin V, Alwahab UA, Borukh E, Daigle E, Bena J, Pantalone KM, Burguera B. The use of virtual visits for obesity pharmacotherapy in patients with overweight or obesity compared with in-person encounters. Obesity (Silver Spring). 2022 Nov;30(11):2194-2203. doi: 10.1002/oby.23548. Epub 2022 Sep 25. PMID 36156456

RESULTS

PARTICIPANT FLOW:
Groups:
- Virtual Visits: All patients will be seen face to face on visit 1. Patient will be evaluated by an obesity-medicine specialist and also by a registered dietitian and exercise physiologist via telemedicine. Subjects will be prescribed phentermine (37.5 mg po daily; dose may be reduced if not tolerated), and will choose one of two dietary programs (Mediterranean or Keto diet). Weight and vital signs will be monitored remotely and patients will receive a remote scale and a remote blood pressure cuff.
  Subjects will then initiate 3 one to one virtual visits with the obesity specialist. On each of this visit the five pillars of weight management will be discussed including nutrition, physical activity, appetite control, sleep issues, and anxiety/depression/stress. A personalized nutrition and exercise program will be developed. If felt relevant by the provider, subjects may also be referred to a mental health specialist and/or sleep clinic. All medical care will be provided virtually.
  Phentermine 37.5 Mg: Patients will receive 37.5 mg of phentermine daily for a 12 week duration
  Dietary program: Patients will be able to select either the Mediterranean diet or the Ketogenic diet and will work with a dietician
  Exercise program: Patients will be provided with a personalized exercise program
- Face to Face Visits: All patients independently of the randomization arm will be seen face to face on visit 1. Patients will be evaluated by an obesity-medicine specialist and patient will also be seen face to face by a registered dietitian and exercise physiologist. Subjects will be prescribed phentermine (37.5 mg po daily; dose may be reduced if not tolerated). Patients will choose one of two dietary programs (Mediterranean or Keto diet). Weight and vital signs will be monitored in each of the visits.
  Subjects will then initiate 3 face to face visits with the obesity specialist provider every 4 weeks. The five pillars of weight management will be discussed including nutrition, physical activity, appetite control, sleep issues, and anxiety/depression/stress.
  The patient will be provided a personalized nutrition and exercise program and may be referred to a mental health specialist and/or sleep clinic per provider discretion. All medical care will be provided via a face-to-face manner.
  Phentermine 37.5 Mg: Patients will receive 37.5 mg of phentermine daily for a 12 week duration
  Dietary program: Patients will be able to select either the Mediterranean diet or the Ketogenic diet and will work with a dietician
  Exercise program: Patients will be provided with a personalized exercise program
Period: Overall Study
Arm/Group | Virtual Visits | Face to Face Visits
Started | 35 | 35
Completed | 32 | 32
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Visits | Face to Face Visits | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 35 | 70
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 63
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 30 | 35 | 65
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 19 | 31
  White | 19 | 14 | 33
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight (Percentage)
Description: The primary endpoint is mean change in body weight (%) from baseline (visit 1) to 12 weeks (visit 4) in body weight.
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: mean change in body weight (%)
Arm/Group | Virtual Visits | Face to Face Visits
Number analyzed (Participants) | 35 | 35
mean change in body weight (%) | -6.61 [-7.72 to -5.49] | -7.68 [-8.9 to -6.45]

2. Secondary Outcome: Adherence to Weight Management Program
Description: Assessed as percentage of patients who completed all visits
Time Frame: 12 weeks
Measure: Number; unit: Percentage of completed patients
Arm/Group | Virtual Visits | Face to Face Visits
Number analyzed (Participants) | 35 | 35
Percentage of completed patients | 82.9 | 62.9

3. Secondary Outcome: Adherence to Medication Use
Description: Percentage of patients that took the medication as prescribed
Time Frame: 12 weeks
Measure: Number; unit: Percentage of pts completed medication
Arm/Group | Virtual Visits | Face to Face Visits
Number analyzed (Participants) | 35 | 35
Percentage of pts completed medication | 93.3 | 83.3

4. Secondary Outcome: Percentage of Patients That Tolerated Full Dosage of Phentermine (37.5mg)
Time Frame: 12 weeks
Measure: Number; unit: Percentage of patients on full dose
Arm/Group | Virtual Visits | Face to Face Visits
Number analyzed (Participants) | 35 | 35
Percentage of patients on full dose | 85.7 | 90

5. Secondary Outcome: Percentage of Patients Who Achieved More Than 5% Weight Loss Over the Course of the Study (12 Weeks)
Time Frame: 12 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of patients with >5% wt loss
Arm/Group | Virtual Visits | Face to Face Visits
Number analyzed (Participants) | 35 | 35
Percentage of patients with >5% wt loss | 64.7 [50.5 to 82.9] | 70.5 [55.1 to 90.1]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 12 weeks
Arm/Group | Virtual Visits | Face to Face Visits
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 7/35 | 1/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Virtual Visits (N=35) | Face to Face Visits (N=35)
Nausea/Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Right paresthesia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness/fainting (Nervous system disorders) | 1 (1) | 0 (0)
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wrist Strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT04614545/Prot_SAP_000.pdf